CLINICAL TRIAL: NCT03341689
Title: Safety and Efficacy of Psilocybin for the Treatment of Headache Disorders: Sub-Study I
Brief Title: Psilocybin for the Treatment of Migraine Headache
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Ceruvia Lifesciences (Unknown)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1607018057.A
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Migraine Headache
Keywords: Psilocybin
MeSH Terms: conditions — Migraine Disorders | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo/Low Dose Psilocybin (Experimental): Subjects in this arm receive placebo in the first session and low dose psilocybin in the second session.
  Interventions: Drug: Low Dose Psilocybin; Drug: Placebo
- Placebo/High Dose Psilocybin (Experimental): Subjects in this arm receive placebo in the first session and high dose psilocybin in the second session.
  Interventions: Drug: High Dose Psilocybin; Drug: Placebo
- Low Dose Psilocybin/Placebo (Experimental): Subjects in this arm receive low dose psilocybin in the first session and placebo in the second session.
  Interventions: Drug: Low Dose Psilocybin; Drug: Placebo
- High Dose Psilocybin/Placebo (Experimental): Subjects in this arm receive high dose psilocybin in the first session and placebo in the second session.
  Interventions: Drug: High Dose Psilocybin; Drug: Placebo

INTERVENTIONS:
Drug: High Dose Psilocybin — 0.143 mg/kg psilocybin capsule
  Arms: High Dose Psilocybin/Placebo; Placebo/High Dose Psilocybin
Drug: Low Dose Psilocybin — 0.0143 mg/kg psilocybin capsule
  Arms: Low Dose Psilocybin/Placebo; Placebo/Low Dose Psilocybin
Drug: Placebo — microcrystalline cellulose capsule

SUMMARY:
The purpose of this study is to investigate the effects of oral psilocybin in migraine headache. Subjects will each receive a dose of placebo and a dose of psilocybin approximately 14 days apart. Subjects will be randomized to the order of treatment and they will be randomized to receive either low or high dose psilocybin. Subjects will maintain a headache diary prior to, during, and after the treatments in order to document headache frequency and intensity, as well as associated symptoms. This preliminary study will inform on the basic effects of psilocybin in migraine headache and inform on the design of larger, more definitive studies.

DETAILED DESCRIPTION:
The number of arms reflects the design of the enhanced blinding method. The final enrollment number reflects the number of subjects participating in study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine headache per ICHD-3beta criteria
* Typical pattern of migraine attacks with approximately two migraines or more weekly
* Attacks are managed by means involving no more than twice weekly triptan use
* Age 21 to 65

Exclusion Criteria:

* Axis I psychotic disorder (e.g. schizophrenia, bipolar I, depression with psychosis)
* Axis I psychotic disorder in first degree relative
* Unstable medical condition, severe renal, cardiac or hepatic disease, pacemaker, or serious central nervous system pathology
* Pregnant, breastfeeding, lack of adequate birth control
* History of intolerance to psilocybin, LSD, or related compounds
* Drug or alcohol abuse within the past 3 months (excluding tobacco)
* Urine toxicology positive to drugs of abuse
* Use of vasoconstrictive medications (i.e. sumatriptan, pseudoephedrine, midodrine) within 5 half-lives of test days
* Use of serotonergic antiemetics (i.e. ondansetron) in the past 2 weeks
* Use of antidepressant medication (i.e. TCA, MAOI, SSRI) in the past 6 weeks
* Use of steroids or certain other immunomodulatory agents (i.e. azathioprine) in the past 2 weeks

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change in migraine headache days | From two weeks before first session to two weeks after second session using a headache diary
  Average days (number of days per week)
Change in migraine attack frequency | From two weeks before first session to two weeks after second session using a headache diary
  Average number (number per week)
Change in migraine attack duration | From two weeks before first session to two weeks after second session using a headache diary
  Average duration (measured in hours)
Change in pain intensity of migraine attacks | From two weeks before first session to two weeks after second session using a headache diary
  Average pain intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of nausea/vomiting during migraine attacks | From two weeks before first session to two weeks after second session using a headache diary
  Average intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of photophobia | From two weeks before first session to two weeks after second session using a headache diary
  Average intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of phonophobia | From two weeks before first session to two weeks after second session using a headache diary
  Average intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in migraine attack-related functional disability | From two weeks before first session to two weeks after second session using a headache diary
  Average disability (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)

SECONDARY OUTCOMES:
Change in the use of abortive/rescue medication | From two weeks before first session to two weeks after second session using a headache diary
  number of days (number of days per week using a migraine abortive)
Time to first migraine attack | From the day of each session until two weeks after each test session
  Measured in days
Time to second migraine attack | From the day of each session until two weeks after each test session
  Measured in days
Quality of life using the Centers for Disease Control (CDC) Health-Related Quality of Life Scale: Healthy Days Symptoms Module | From two weeks before first session to three months after second session using a headache diary
  4 questions scored 0 to 30 each; higher numbers indicate worse quality of life.
  (1) pain-related impairment, (2) mood symptoms, (3) anxiety symptoms, and (4) lack of sleep Percent change for each measure as well as total score (range 0 to 120) will be calculated.
Psychedelic effects using the 5-Dimensional Altered States of Consciousness (5D-ASC) scale | Taken on each test day approximately 6 hours after drug administration
  94 questions scored 0 to 100 each; higher numbers indicate greater psychedelic effects Questions address 5 dimensions: (1) Oceanic boundlessness (score range 0-2700), (2) Dread of Ego Dissolution (score range 0-2100), (3) Visionary Restructuralization (score range 0-1800), (4) Auditory Alterations (score range 0-1600), and (5) Vigilance reduction (score range 0-1200) Score for each dimension as well as total score (range 0 to 9400) will be measured.
Change in blood pressure | Measured during each test session prior to drug administration, every 15 minutes in the first hour, every 30 minutes in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change in mean arterial blood pressure from baseline during each test day (mmHg)
Change in heart rate | Measured during each test session prior to drug administration, every 15 min in the first hour, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each test day (beats per minute)
Change in peripheral oxygenation | Measured during each test session prior to drug administration, every 15 min in the first hour, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each test day (SpO2)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven Campus, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Schindler EAD, Sewell RA, Gottschalk CH, Luddy C, Flynn LT, Lindsey H, Pittman BP, Cozzi NV, D'Souza DC. Exploratory Controlled Study of the Migraine-Suppressing Effects of Psilocybin. Neurotherapeutics. 2021 Jan;18(1):534-543. doi: 10.1007/s13311-020-00962-y. Epub 2020 Nov 12. PMID 33184743